CLINICAL TRIAL: NCT04901195
Title: A Phase 3, Open-Label, Parallel Group, Multicenter, Extension Study Evaluating the Long-Term Treatment of Bimekizumab in Study Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Test the Long-term Treatment of Bimekizumab in Study Participants With Moderate to Severe Hidradenitis Suppurativa
Acronym: BE HEARD EXT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS0005; 2020-004179-42 (EudraCT Number); U1111-1307-6132 (Other: World Health Organization (WHO)); 2024-511035-10 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: Bimekizumab; UCB4940; HS; Hidradenitis Suppurativa; Acne inversa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab dosing regimen 1 (Experimental): Subjects participating in the study will receive assigned bimekizumab dosing regimen 1 during the open-label extension period.
  Interventions: Drug: Bimekizumab
- Bimekizumab dosing regimen 2 (Experimental): Subjects participating in the study will receive assigned bimekizumab dosing regimen 2 during the open-label extension period.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: UCB4940

SUMMARY:
The purpose of the study is to evaluate the safety of long-term therapy of bimekizumab in study participants with moderate to severe hidradenitis suppurativa (HS)

ELIGIBILITY:
Inclusion Criteria:

* Study participant has completed the Maintenance Treatment Period through Week 48 in HS0003 (NCT04242446) or HS0004 (NCT04242498), was eligible to receive bimekizumab at the time of completing the feeder study, and did not meet any withdrawal criteria of the feeder study
* Study participant is considered reliable and capable of adhering to the protocol (eg, able to understand and complete questionnaires), visit schedule, and medication intake according to the judgement of the Investigator
* A female study participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the contraceptive guidance during the open-label extension period and for at least 20 weeks after the final dose of investigational medicinal product (IMP)

Exclusion Criteria:

* Female study participant who is breastfeeding, pregnant, or plans to become pregnant during the study or within 20 weeks following the final dose of investigational medicinal product (IMP)
* Study participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the participant's ability to participate in this study as determined by the Investigator based on protocol required assessments Note: For any study participant with an ongoing serious adverse event (SAE) from HS0003 (NCT04242446) or HS0004 (NCT04242498), or any current sign or symptom that may indicate a medically significant active infection (except for the common cold) or has had an infection requiring systemic antibiotics within 2 weeks of study entry or a history of serious infections in HS0003 or HS0004, the Medical Monitor must be consulted prior to the study participant's entry into HS0005, although the decision on whether to enroll the participant remains with the Investigator.
* Study participant has a positive or indeterminate interferon-gamma release assay (IGRA) in a feeder study, unless appropriately evaluated and treated
* Study participant has ongoing or planned use of prohibited hidradenitis suppurativa (HS) or non-HS treatment
* Study participant plans to participate in another study of a medicinal product or device under investigation during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events (TEAEs) during the study | From Baseline (Day 1) until end of Safety Follow-Up (up to Week 196)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP.

SECONDARY OUTCOMES:
Percentage of participants with treatment-emergent serious adverse events (SAEs) during the study | From Baseline (Day 1) until end of Safety Follow-Up (up to Week 196)
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical events
Percentage of participants with treatment-emergent adverse events (TEAEs) leading to withdrawal from the study | From Baseline (Day 1) until end of Safety Follow-Up (up to Week 196)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs leading to discontinuation of the study are reported.
Percentage of participants achieving clinical response as measured by Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) | Week 0, Week 16, Week 32, Week 48, Week 76, Week 92, Week 100, Week 116, Week 132, Week 148, Week 164, and Week 180
  HiSCR50 is defined as at least a 50 % reduction from Baseline in the total abscess and inflammatory nodule (AN) count, with no increase from Baseline in abscess or draining tunnel count.
  Results will be presented individually per week listed under time points.
Percentage of participants achieving clinical response as measured by Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) | Week 0, Week 16, Week 32, Week 48, Week 76, Week 92, Week 100, Week 116, Week 132, Week 148, Week 164, and Week 180
  HiSCR75 is defined as at least a 75 % reduction from Baseline in the total abscess and inflammatory nodule (AN) count, with no increase from Baseline in abscess or draining tunnel count.
  Results will be presented individually per week listed under time points.
Percentage of participants with Flare | Week 0, Week 16, Week 32, Week 48, Week 76, Week 92, Week 100, Week 116, Week 132, Week 148, Week 164, and Week 180
  Flare is defined as a ≥25 % increase in abscess and inflammatory nodule (AN) count with an absolute increase in AN count of ≥2 relative to Baseline.
  Results will be presented individually per week listed under time points.
Hidradenitis Suppurativa Symptom Questionnaire (HSSQ) Response for Worst Pain | Week 0, Week 16, Week 32, Week 48, Week 76, Week 92, Week 100, Week 116, Week 132, Week 148, Week 164, and Week 180
  The 4 items on the HSSQ assess the study participant's perception of the core symptoms of HS experienced in the past 7 days - pain, smell or odor, drainage or oozing from HS lesions, and itch on an 11-point numeric rating scale with higher scores indicating higher symptom level.
  Results will be presented individually per week listed under time points.
Absolute change from Baseline in Dermatology Life Quality Index (DLQI) Total Score | Week 0, Week 16, Week 32, Week 48, Week 76, Week 92, Week 100, Week 116, Week 132, Week 148, Week 164, and Week 180
  The DLQI is a skin disease specific questionnaire aimed at the evaluation of how the disease affects participants health related quality of life (QOL). The DLQI total score ranges from 0 to 30 with higher scores indicating higher skin disease impact on QOL.
  Results will be presented individually per week listed under time points.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (145):
- United States (43):
  - Hs0005 50140, Birmingham, Alabama
  - Hs0005 50175, Phoenix, Arizona
  - Hs0005 50162, Fountain Valley, California
  - Hs0005 50161, Los Angeles, California
  - Hs0005 50220, San Diego, California
  - Hs0005 50196, Thousand Oaks, California
  - Hs0005 50199, Miami, Florida
  - Hs0005 50205, North Miami Beach, Florida
  - Hs0005 50152, Orange Park, Florida
  - Hs0005 50184, Pembroke Pines, Florida
  - Hs0005 50193, Sandy Springs, Georgia
  - Hs0005 50280, Watkinsville, Georgia
  - Hs0005 50234, Plainfield, Indiana
  - Hs0005 50425, Murray, Kentucky
  - Hs0005 50198, Beverly, Massachusetts
  - Hs0005 50146, Boston, Massachusetts
  - Hs0005 50178, Clarkston, Michigan
  - Hs0005 50105, St Louis, Missouri
  - Hs0005 50194, Omaha, Nebraska
  - Hs0005 50208, Las Vegas, Nevada
  - Hs0005 50159, Newington, New Hampshire
  - Hs0005 50137, East Windsor, New Jersey
  - Hs0005 50200, Verona, New Jersey
  - Hs0005 50237, Albuquerque, New Mexico
  - Hs0005 50235, New York, New York
  - Hs0005 50151, Chapel Hill, North Carolina
  - Hs0005 50211, Durham, North Carolina
  - Hs0005 50179, Winston-Salem, North Carolina
  - Hs0005 50177, Cincinnati, Ohio
  - Hs0005 50138, Columbus, Ohio
  - Hs0005 50145, Columbus, Ohio
  - Hs0005 50202, Fairborn, Ohio
  - Hs0005 50204, Tulsa, Oklahoma
  - Hs0005 50147, Hershey, Pennsylvania
  - Hs0005 50008, Johnston, Rhode Island
  - Hs0005 50180, Providence, Rhode Island
  - Hs0005 50084, Charleston, South Carolina
  - Hs0005 50236, Greenville, South Carolina
  - Hs0005 50142, Nashville, Tennessee
  - Hs0005 50201, Arlington, Texas
  - Hs0005 50148, Pflugerville, Texas
  - Hs0005 50141, Salt Lake City, Utah
  - Hs0005 50270, Seattle, Washington
- Australia (8):
  - Hs0005 30015, Campbelltown
  - Hs0005 30016, Carlton
  - Hs0005 30011, East Melbourne
  - Hs0005 30017, Kogarah
  - Hs0005 30018, Parkville
  - Hs0005 30014, St Leonards
  - Hs0005 30009, Westmead
  - Hs0005 30012, Woolloongabba
- Belgium (2):
  - Hs0005 40002, Leuven
  - Hs0005 40121, Woluwe-Saint-Lambert
- Bulgaria (6):
  - Hs0005 40313, Pleven
  - Hs0005 40284, Sofia
  - Hs0005 40311, Sofia
  - Hs0005 40314, Sofia
  - Hs0005 40315, Sofia
  - Hs0005 40353, Stara Zagora
- Canada (9):
  - Hs0005 50233, Barrie
  - Hs0005 50172, Cobourg
  - Hs0005 50135, Edmonton
  - Hs0005 50174, London
  - Hs0005 50190, Richmond Hill
  - Hs0005 50192, Saskatoon
  - Hs0005 50133, Surrey
  - Hs0005 50134, Waterloo
  - Hs0005 50136, Winnipeg
- Czechia (2):
  - Hs0005 40063, Prague
  - Hs0005 40194, Prague
- France (14):
  - Hs0005 40197, Amiens
  - Hs0005 40245, Antony
  - Hs0005 40321, Auxerre
  - Hs0005 40320, La Rochelle
  - Hs0005 40355, Le Mans
  - Hs0005 40247, Lyon
  - Hs0005 40130, Marseille
  - Hs0005 40132, Nice
  - Hs0005 40404, Reims
  - Hs0005 40318, Rouen
  - Hs0005 40403, Saint-Etienne
  - Hs0005 40246, Saint-Mandé
  - Hs0005 40285, Toulon
  - Hs0005 40286, Toulouse
- Germany (15):
  - Hs0005 40325, Berlin
  - Hs0005 40326, Berlin
  - Hs0005 40248, Bochum
  - Hs0005 40327, Bonn
  - Hs0005 40288, Darmstadt
  - Hs0005 40324, Dresden
  - Hs0005 40356, Dresden
  - Hs0005 40287, Frankfurt am Main
  - Hs0005 40142, Hamburg
  - Hs0005 40328, Hanover
  - Hs0005 40249, Kiel
  - Hs0005 40250, Lübeck
  - Hs0005 40174, Mainz
  - Hs0005 40323, München
  - Hs0005 40177, Münster
- Greece (2):
  - Hs0005 40251, Athens
  - Hs0005 40252, Efkarpia
- Hs0005 40254, Debrecen, Hungary
- Hs0005 40344, Dublin, Ireland
- Italy (4):
  - Hs0005 40261, Catania
  - Hs0005 40263, Roma
  - Hs0005 40258, Rozzano
  - Hs0005 40330, Torino
- Japan (13):
  - Hs0005 20196, Bunkyō City
  - Hs0005 20144, Fukuoka
  - Hs0005 20043, Itabashi-ku
  - Hs0005 20195, Kagoshima
  - Hs0005 20170, Kurume
  - Hs0005 20190, Kyoto
  - Hs0005 20033, Nagoya
  - Hs0005 20152, Nakagami-gun
  - Hs0005 20178, Nishinomiya
  - Hs0005 20153, Obihiro
  - Hs0005 20037, Osaka
  - Hs0005 20154, Sapporo
  - Hs0005 20171, Sendai
- Netherlands (3):
  - Hs0005 40351, Breda
  - Hs0005 40292, Groningen
  - Hs0005 40264, Rotterdam
- Poland (6):
  - Hs0005 40347, Lodz
  - Hs0005 40293, Rzeszów
  - Hs0005 40335, Warsaw
  - Hs0005 40095, Wroclaw
  - Hs0005 40333, Wroclaw
  - Hs0005 40334, Wroclaw
- Spain (10):
  - Hs0005 40266, Badalona
  - Hs0005 40159, Barcelona
  - Hs0005 40267, Barcelona
  - Hs0005 40298, Granada
  - Hs0005 40294, Las Palmas de Gran Canaria
  - Hs0005 40268, Madrid
  - Hs0005 40297, Manises
  - Hs0005 40295, Pontevedra
  - Hs0005 40049, Seville
  - Hs0005 40230, Valencia
- Hs0005 40406, Geneva, Switzerland
- Turkey (Türkiye) (4):
  - Hs0005 40270, Antalya
  - Hs0005 40273, Gaziantep
  - Hs0005 40272, Istanbul
  - Hs0005 40271, Izmir
- Hs0005 40339, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Derived] Skrzypczak T, Skrzypczak A, Matusiak L, Szepietowski JC. An evaluation of bimekizumab for the treatment of hidradenitis suppurativa. Expert Opin Biol Ther. 2025 Aug;25(8):811-819. doi: 10.1080/14712598.2025.2522119. Epub 2025 Jun 21. PMID 40524676